CLINICAL TRIAL: NCT05920408
Title: A Phase 1B/2A Study to Assess the Safety, Tolerability, Pharmacokinetic and Anti-tumoral Activity of EXS21546 in Combination With a PD-1 Inhibitor in Patients With Advanced Solid Tumours
Brief Title: Study to Assess EXS21546 in Combination in Patients With Advanced Solid Tumours
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Emerging data demonstrates challenge for EXS21546 to reach suitable therapeutic index.
Sponsor: Exscientia AI Limited (Industry)
Collaborators: Biotrial (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EXS21546-002
Record Dates: First submitted 2023-05-18; First posted 2023-06-27 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Advanced Solid Tumours

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- EXS21546 (Experimental): EXS21546 Granule in Capsule for oral administration
  Interventions: Drug: EXS21546

INTERVENTIONS:
Drug: EXS21546 — EXS21546 Granule in Capsule

SUMMARY:
A phase 1B/2A study to assess the safety, tolerability, pharmacokinetic and anti-tumoral activity of EXS21546 in combination with a PD-1 inhibitor in patients with advanced solid tumours.

DETAILED DESCRIPTION:
A phase 1B/2A study to assess the safety, tolerability, pharmacokinetic and anti-tumoral activity of EXS21546 in combination with a PD-1 inhibitor, nivolumab, in patients with advanced solid tumours, non small cell lung cancer and renal cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years at time of informed consent.
* Previous histologically confirmed diagnosis of RCC or NSCLC having received previously checkpoint inhibitors as part of a SoC regimen.
* Consent to mandatory paired tumour biopsies of at least one tumour site accessible for repeat biopsies. Planned sites for tumour biopsies must not have been previously irradiated and could be a target lesion of >2 cm diameter according to RECIST v1.1 and must be approved on a case-by-case basis by the Sponsor.
* Measurable disease as per RECIST v1.1 and documented by computed tomography (CT) and/or magnetic resonance imaging (MRI).

Exclusion Criteria:

* Any anti-tumour therapy, including investigational therapies, within 4 weeks prior to the first dose of EXS21546.
* Unresolved or unstable serious toxic side-effects of prior chemotherapy or radiotherapy, i.e., ≥ Grade 2 per CTCAE v5.0.
* Concurrent other malignancy that could interfere with response evaluation.
* Symptomatic central nervous system (CNS) malignancy or metastases. Screening of symptomatic participants without history of CNS metastases is not required. Participants with asymptomatic CNS lesions should have completed standard therapy for their CNS lesions 60 days prior to study enrolment.
* History of interstitial lung disease and/or prior immunotherapy-related pneumonitis.
* Patients who have had or are scheduled to have major surgery < 28 days prior to the first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-04-11 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2023-10-23 (Actual)

PRIMARY OUTCOMES:
Safety of EXS21546 in combination with nivolumab. | Through study completion, an average of 6 months
  Incidence of treatment-emergent adverse events (TEAEs) and SAEs characterised by type, incidence, severity (graded by National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] v5.0), seriousness, timing and relationship to EXS21546 dosing.
Dose-limiting toxicities (DLTs) of EXS21546 in combination with nivolumab. | Through dose escalation completion, an average of 6 months
  Incidence of dose limiting toxicities (DLTs) during Cycle 1 (initial 28 days) of treatment with escalating doses of EXS21546 in combination with an approved dose of nivolumab.
Preliminary anti-tumoural activity of EXS21546 in combination with nivolumab. | Through study completion, an average of 6 months
  Objective response rate (ORR) per Response Evaluation Criteria in Solid Tumours (RECIST) v1.1.
Treatment adherence of EXS21546 in combination with nivolumab. | Through study completion, an average of 6 months
  Number of doses recorded in the treatment diary.
Tolerability of EXS21546 in combination with nivolumab. | Through study completion, an average of 6 months
  Frequency of dose interruptions, dose reductions and dose intensity achieved.

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Italiano, MD, Principal Investigator — Institut Bergonie, Bordeaux, France
Locations (5):
- Belgium (2):
  - Institute Jules Bordet, Brussels
  - CHU Mont-Godinne, Namur
- France (3):
  - Institut Bergonie, Bordeaux
  - Centre GF Leclerc, Dijon
  - Centre Eugene Marquis, Rennes

IPD SHARING:
Plan to Share IPD: No